CLINICAL TRIAL: NCT02753049
Title: Adherence Connection for Counseling, Education, and Support (ACCESS): A Proof of Concept Study
Brief Title: Adherence Connection for Counseling, Education, and Support
Acronym: ACCESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Ann-Margaret Dunn Navarra, Assistant Professor, New York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1K23NR015970-02 (NIH)
Record Dates: First submitted 2016-04-08; First posted 2016-04-27 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: HIV-infection/AIDS
Keywords: HIV; AIDS; Adolescent; Adherence; Retention; mHealth
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Peer led mHealth adherence intervention (Experimental): Eligible participants enrolled will receive five, weekly-60 minute, 'ACCESS' sessions, delivered by a peer adherence coach via remote videoconferencing, using smartphones. Cognitive behavioral strategies will be employed to target beliefs about antiretroviral treatment (ART), knowledge of ART, and adherence self-efficacy.
  Interventions: Behavioral: Peer led mHelath behavioral intervention

INTERVENTIONS:
Behavioral: Peer led mHelath behavioral intervention — A trained peer adherence coach will schedule five, weekly-60 minute, 'ACCESS' sessions, delivered to participants via remote videoconferencing, using smartphones. Cognitive behavioral strategies will be employed to target beliefs about antiretroviral treatment (ART), knowledge of ART, and adherence self-efficacy.
  Other Names: ACCESS

SUMMARY:
This Mentored Patient-Oriented Research Career Development Award - (K23) seeks to provide the advanced knowledge, skills, and experience for the candidate's career transition to an independent nurse scientist. Her long term goal is to become a leading nurse scientist in designing, implementing, and evaluating technology supported behavioral interventions targeted for improved disease self-management (i.e. medication adherence, retention in care) among human immunodeficiency virus (HIV)-infected, ethnic minority adolescents and young adults. With an extensive background in pediatric HIV nursing and completed NIH funded pre and post-doctoral interdisciplinary research traineeships, the candidate has begun to develop the knowledge-base and skills necessary for this goal.

This award details a 3-year scope of mentored career development through which she will gain the foundation for future research endeavors. Specifically, the goals of this proposal are to: 1) conduct a novel research project under the mentorship of an interdisciplinary team of expert researchers; 2) acquire expertise in health informatics for implementation of technology supported behavioral interventions, health disparities, and advanced qualitative and mixed methods design and analysis through firsthand experience, didactic interactions with mentors, and graduate level coursework; 3) build a network of colleagues and collaborators within New York University and elsewhere through this research and participation at national and international meetings; and 4) prepare and submit a federal research grant (R-21) based upon the skills and findings from this award period.

The specific research project through which she will accomplish these goals is a proof of concept study, Adherence Connection for Counseling, Education, and Support (ACCESS), and addresses the challenge of adherence to antiretroviral treatment among HIV-infected adolescents and young adults. A mixed method design is proposed and the specific aims are to: 1) Characterize the feasibility and acceptability of a peer led, mHealth cognitive behavioral intervention delivered via remote videoconferencing using smartphones; 2) Obtain initial estimates of the biobehavioral impact of ACCESS on HIV virologic outcomes and self-reported ART adherence, beliefs and knowledge about antiretroviral treatment, adherence self-efficacy, and healthcare utilization (retention in HIV care). In summary, the ACCESS adherence intervention is consistent with the National Institute of Nursing Research (NINR) call for the development of novel interventions to deliver personalized care and real-time health information for patients.

ELIGIBILITY:
1. HIV seropositive status (perinatally and behaviorally infected youth)
2. Ages 16-29 years
3. English speaking
4. Current ART with a prescribed regimen
5. Evidence of virologic failure or (detectable quantitative HIV serum viral load>200 copies/ml)
6. No neuro-cognitive deficits which would impede participation in videoconferencing sessions or completion of study measures. [Screening with the Folstein Mini-Mental State Exam (MMSE) will be performed to assess for the presence of neurocognitive deficits. Participants with a score of 24 or greater will be eligible for study participation.]

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-23 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Change in Serum HIV RNA quantitative viral load | Serum HIV RNA quantitative viral load will be measured at baseline and at 8 weeks, 16 weeks, and 24 weeks post-intervention.
  Serum HIV RNA quantitative viral load results will be available for medical record data extraction at four time points, baseline (pre-intervention), and weeks 8, 16 & 24 post-intervention. The primary outcome variable of adherence as measured with serum HIV-RNA will be dichotomized as a binary variable (< 48 copies/ml; > 48 copies/ml), indicating viral suppression. An interval estimate of the odds ratio will indicate the potential impact of ACCESS on viral suppression, with Chi-Square or Fisher's Exact Test for statistical significance.

OTHER OUTCOMES:
Change in Beliefs about antiretroviral treatment | Beliefs about antiretroviral treatment will be measured at baseline and 24 weeks.
  Beliefs about ART will be assessed with the Beliefs about Medication Scale (BAMS)- a 59 item health beliefs questionnaire using a 7-point Likert scale to assess perceived threat, positive outcome expectancy, negative outcome expectancy, and intent regarding oral medication adherence [Riekert K. et al. 2002; J Clinical Psychol Med Settings]. Changes in scores of beliefs about medications will be compared pre and post the ACCESS intervention using Chi-Square or Fisher's Exact Test for discrete variables, and paired t-tests for continuous variables.
Change in Knowledge about antiretroviral treatment | Knowledge about antiretroviral therapy will be measured at baseline and 24 weeks.
  Knowledge about antiretroviral treatment will be measured with the HIV Treatment Knowledge Scale. This 21 item instrument uses true and false questions to assess knowledge of adherence, side effects and antiretroviral resistance [Balfour L. et al. 2007; AIDS Care]. Changes in scores of knowledge about ART will be compared pre and post the ACCESS intervention using Chi-Square or Fisher's Exact Test for discrete variables, and paired t-tests for continuous variables.
Change in Adherence Self-Efficacy | Adherence self-efficacy will be measured at baseline and 24 weeks.
  Adherence self-efficacy will be measured with the Adherence Self-Efficacy Scale - a 12 item survey measure that uses a 10 point scale (0=cannot do it all;10=completely certain can do it) to assess confidence in ability to carry out important treatment related behaviors [Johnson M. et al. 2007; J Behav Med].
  Changes in scores of self-efficacy will be compared pre and post the ACCESS intervention using Chi-Square or Fisher's Exact Test for discrete variables, and paired t-tests for continuous variables.
Change in 3-day adherence estimate | 3-day adherence estimates will be measured at baseline, and 8 weeks, 16 weeks, and 24 weeks
  An average missed dose calculation will be computed and operationalized as: # of doses missed per medication multiplied by dosing schedule during the past 3 days/ divided by total number of prescribed doses over past 3 days. This percentage will be subtracted from 100% to obtain the 3-day adherence estimate [Garvie P. et al. 2010; J Adol Health]
Change in health care utilization (retention in care) | Retention in care will be measured at baseline and 24 weeks
  For the purposes of this proof of concept study, retention in HIV care will be calculated as a proportion of kept to scheduled visits (range 0-100%). Changes in scores of healthcare utilization (retention) will be compared pre and post the ACCESS intervention using Chi-Square or Fisher's Exact Test for discrete variables, and paired t-tests for continuous variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Bellevue Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided